CLINICAL TRIAL: NCT04284046
Title: CT Scores Predict Mortality in 2019-nCoV Pneumonia
Status: Completed | Type: Observational
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ruilan Wang, PhD, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: CT2019-nCoV
Record Dates: First submitted 2020-02-22; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: CT Scores Predict Mortality in 2019-nCoV Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High CT score
  Interventions: Other: CT score
- Low CTscore
  Interventions: Other: CT score

INTERVENTIONS:
Other: CT score — CT score = normal lung tissue (%) ×1 + GGO (%) ×2 + consolidation (%) ×3

SUMMARY:
While 2019-nCoV nucleic acid swab tests has high false positives rate, How to diagnose 2019-nCoV pneumonia and predict prognosis by CT is very important.In this retrospective single-center study, we consecutively included suspected 2019-nCoV pneumonia critical cases in the intensive care unit of Wuhan third hospital from January 31, 2020 to February 16, 2020. The cases were confirmed by real-time RT-PCR, and all patients were evaluated with CT, cutoff values were obtained according to the Yoden index, and were divided into high CT score group and low CT score group. Epidemiological, demographic, clinical, and laboratory data were collected.

ELIGIBILITY:
Inclusion Criteria:

* all patients suspected of 2019 novel coronavirus infection.

Exclusion Criteria:

* patients' data are not available.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients suspected of 2019 novel coronavirus infection.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
7-day mortality | 7-day

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan third hospital, Wuhan, Hubei, China